CLINICAL TRIAL: NCT05095883
Title: Correlation Between Body Weight and Foot Progression Angle in Adolescents
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant. Professor of physical therapy, Department of Physical Therapy for Pediatrics, Delta University for Science and Technology
Other Study IDs: adolecents foot angles
Record Dates: First submitted 2021-09-17; First posted 2021-10-27 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Adolescent; Adolescent Development
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy: Children in this group will be healthy category according to CDC chart which ranged from BMI-for-age 5th to 85th percentiles
- overweight: Children in this group will be overweight category according to CDC chart which ranged from BMI-for-age 85th to 95th percentiles
- obese: Children in this group will be obese category according to CDC chart which ranged from BMI-for-age > 95th percentiles
- underweight: Children in this group will be underweight category according to CDC chart ranged from BMI-for-age < 5th percentiles

SUMMARY:
Obesity is associated with functional decline , altered spatiotemporal gait parameters (e.g. lower gait speed, shorter strides, and increased step width), and a significantly higher metabolic cost of walking compared to people with normal body weight. Obesity also negatively affects balance control.This study will investigate foot progression angle in adolescents related to their weight and category classification based on the CDC (Centers for Disease Control and Prevention) growth charts.

ELIGIBILITY:
Inclusion Criteria:

* All children have normal stature for age percentile according to CDC chart.
* The sample will include both sex and will be divided in to 4 groups according to the CDC (Centers for Disease Control and Prevention) growth charts.
* All children are normal &perform all activities of daily living
* They were able to understand and follow verbal commands and instructions included in the testing procedures.

Exclusion criteria:

* All of them could be part of recreational activities in their public schools but no competitive sports. Children who participated in any regular sport activities involving the lower extremities will be excluded.
* None of them had any surgical intervention in the lower extremities.
* None of them had any history of musculoskeletal deformities or neuromuscular disorders.
* They had neither visual, auditory defect.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Two hundred healthy non-athletic children from both sexes will participate in this study.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
foot progression angle for healthy group | assessed immediately after the procedure
  participants in healthy group will be assessed for foot progression angle (FPA). The FPA is defined as the angle made by the long axis of the foot from the heel to 2nd metatarsal and the line of progression of gait
foot progression angle for overweight group | assessed immediately after the procedure
  participants in overweight group will be assessed for foot progression angle (FPA). The FPA is defined as the angle made by the long axis of the foot from the heel to 2nd metatarsal and the line of progression of gait.
foot progression angle for obese group | assessed immediately after the procedure
  participants in obese group will be assessed for foot progression angle (FPA). The FPA is defined as the angle made by the long axis of the foot from the heel to 2nd metatarsal and the line of progression of gait.
foot progression angle for underweight group | assessed immediately after the procedure
  participants in underweight group will be assessed for foot progression angle (FPA). The FPA is defined as the angle made by the long axis of the foot from the heel to 2nd metatarsal and the line of progression of gait.

CONTACTS AND LOCATIONS:
Locations (1):
- AAA, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided